CLINICAL TRIAL: NCT02608151
Title: Effect in the Short and Medium Term of Different Techniques of Tactile Stimulations on Neurological Development in a Population of Very Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011-08; RC12_3135 (Other: APHM)
Record Dates: First submitted 2015-10-22; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Very Preterm Infant
Keywords: neurodevelopement; Very preterm infant
MeSH Terms: interventions — Massage; Oils

ARMS (2):
- Touch massage without oil (Active Comparator): massage without oil
  Interventions: Other: massage without oil
- touch massage with oil (Experimental): massage with an oil consisting of 4 vegetable oils (40% sunflower oil, 3% grape seed oil, 1.5% coriander oil, and 57% of rapeseed oil)
  Interventions: Other: massage with oil

INTERVENTIONS:
Other: massage with oil — Application or not of an oil consisting of 4 vegetable oils (40% sunflower oil, 3% grape seed oil, 1.5% coriander oil, and 57% of rapeseed oil) during the massage. This oil was chosen due to its composition of essential fatty acids (60%) including: linoleic acid (omega 6,25g 100 g)), linolenic acid (omega 3 5.3g to 100 g) and tocopherol (vitamin E) .
  Arms: touch massage with oil
Other: massage without oil
  Arms: Touch massage without oil

SUMMARY:
Premature birth deprives infants of sensory stimulation. Tactile stimulation such as massage pressure with kinesthetic movement significantly increases the weight, bone density and shorten the duration of stay of premature babies who benefits.

Studies using vegetable oils show an increase in the effect on weight gain by cutaneous absorption. The mechanism is probably vagal (stimulation of baroreceptors and skin mechanoreceptors) since it is found in children stimulated an increase in the vagal activity, acceleration of gastric emptying and an increase in the secretion of insulin and IGF1.

Few studies have evaluated the effects of massage on the medium-term neurological development in preterm infants and the effect of the essential oils in the effectiveness of touching the short and medium term massage.

The aim of the investigators study is to evaluate the neurological development in the short and medium term in premature newborns and biological effects of massage with essential use of vegetable oil.

Methodology and possible collaborations This is a monocentric, randomized, controlled, in a neonatal intensive care unit. It concerns 60 children born between 26 and 30 weeks of amenorrhea. Each child receives massage randomized with or without oil ISIO 4. The treatment is administered 10 minutes twice a day for 10 consecutive days watching for signs of intolerance. The quality of the spontaneous motility between 12 and 20 weeks of age corrected is used as the first neurological assessment criterion.

The questionnaire (ASQ) Bricker and Squires (translated into French by Martha Bonin et al.) is used to 6, 12, 24 months corrected age and completed by the parents as a second neurological endpoint.

A lipid chromatography is performed at the beginning and at the end of the massage time and at the deliverance from NICU for comparing the profile of children's fatty acids.

Expected results Show that there is an improvement in the neurological development in children who received massage with vegetable oil ISIO 4. Show that there is a skin absorption of essential fatty acids that can substitute for a known major deficiency in premature even in infants fed breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Children whose term of birth is between 26 and 31 weeks of amennorhea
* Children's age less than or equal to 33 weeks of postnatal age
* Children without neurological pathologies (intra ventricular hemorrhage grade 1 or 2 of the papilla transfontanellar ultrasound [Papille 1978] and / or brain abnormalities on MRI type of 1-4 according to modified Paneth classification [Paneth 1999]);
* Children whose parenteral nutrition is less than 60 cc / kg / day;
* Children without infectious disease clinically unstable ( C reactive protein below 7);
* Children without CPAP (Positive Airway Pressure Control) nasal for at least 48 hours;
* Children do not present a genetic syndrome, progressive neurological disease, malformation pathology, a cleft lip and palate;
* Children with one parent or legal representatives are beneficiaries of a social security regimen;

Exclusion Criteria:

* Children under 26 and more than 32 weeks of amenorrhea;
* Children not included at 34 weeks of amenorrhea;
* Children with high-grade intraventricular hemorhage (grade 3-4) [Papille 1978] and / or abnormality of cerebral MRI (grade 5 and 6) [Paneth 1999];
* Children with a necrotizing enterocolitis or nosocomial infection;
* Children with a genetic syndrome, a progressive neurological disease, malformation pathology, a cleft lip and palate.

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Quality of spontaneous movements assessed by motor repertoire score following Prechtl's method | 12-20 weeks post-term
  The primary outcome is represented by the assessment of neuro-development of children from 3 months of age corrected more precisely between 12 and 20 weeks post-term. The evaluation of neuro-development will be realized from measurement of the quality of spontaneous general movement. The motor repertoire was evaluated using the video-recording made between 11 to 16 weeks post-term, following Prechtl's method for the assessment of the motor repertoire between 3 and 5 months. Scores were assigned to the following five aspects: Quality of FMs, Age-adequacy of concurrent movements, Presence and normality of concurrent movements, Presence and normality of postural patterns and Quality of concurrent movements. Scores for each aspect can range from 1 to 4. The scores for the five aspects of the motor repertoire are summed to provide a Motor Optimality Score, range 5 to 20. Higher scores indicate higher movement quality.

SECONDARY OUTCOMES:
Ages and Stages Questionnaire | 3, 6, 12, 18 and 24 months
  The evaluation of neuro-development between 12 and 20 weeks post term from motor score will be complemented by an assessment using the questionnaire "Ages and Stages Questionnaire" (ASQ) at 3, 6, 12, 18 and 24 months. The ASQ [Bricker and Squires 2000] questionnaire is a child developmental delay screening tool, thus identifying children in need of a thorough assessment of their development.
lipid profile | before the procedure (massage program), at the end of the procedure (massage program) and through study completion, an average of 39-40 weeks of amenorrhea corrected age
  The assessment of the lipid profile will be done by analysis of fatty acid profiles of plasma and red blood cells premature by gas chromatography [Ohta 1990].

CONTACTS AND LOCATIONS:
Overall Officials: urielle desalbres, Study Director — APHM
Locations (1):
- APHM, Marseille, France